CLINICAL TRIAL: NCT03339180
Title: Prevalence and Prognostic Implications of Cardiac Injury in Patients With Influenza-like Illness
Brief Title: Cardiac Injury in Patients With Influenza
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anna Nordenskjöld, Principal Investigator, Örebro University, Sweden
Other Study IDs: Do not have any
Record Dates: First submitted 2017-10-26; First posted 2017-11-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Influenza, Human; Myocardial Injury
Keywords: cardiac troponin
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigate the prevalence of elevated biomarkers of cardiac injury in patients with suspected influenza infection and the prognostic implication on the composite endpoint of death of any cause, hospitalization due to myocardial infarction, unstable angina, heart failure and stroke.

DETAILED DESCRIPTION:
The relationship between influenza and cardiovascular events was described in an early study of influenza epidemics from 1915 to 1929 including the 1918-1920 pandemic. Retrospective studies have shown increased risk for acute myocardial infarction (AMI) during the first week following an infection with influenza.

Biochemical markers of cardiac injury such as high sensitive cardiac troponins may be increased during infection with influenza. Increased levels of cardiac troponins are associated with adverse outcome in many different populations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) presenting with influenza-like illness.
* Written informed consent.

Exclusion Criteria:

* Inability to provide informed consent.
* Age <18 years.
* Symptoms indicating an acute coronary syndrome, acute heart failure, rapid atrial fibrillation or acute stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical study will be conducted in Region Örebro County. Recruitment will start October 1st 2017 and is expected to continue for two influenza seasons until April 30, 2019. Individuals for inclusion are recruited among adult patients > 18 years presenting with influenza-like illness at the emergency unit and who, due to strong clinical suspicion of ongoing influenza infection, are tested.
Sampling Method: Probability Sample
Enrollment: 466 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of biochemical markers | One year
  Level of cardiac troponin in patients with influenza The level of hs-cTn, NT-proBNP and hs-CRP at inclusion in patients with and patientes without influenza.
Level of biochemical markers | One year
  Level of other biochemical markers in patients with influenza

SECONDARY OUTCOMES:
Prognostic implication | One year
  Time to all-cause death
Prognostic implication | One year
  Time to admission for myocardial infarction
Prognostic implication | One year
  Time to admission for unstable angina
Prognostic implication | One year
  Time to admission for heart failure
Prognostic implication | One year
  Time to admission for stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided